CLINICAL TRIAL: NCT00264719
Title: Metoclopramide to Aid Establishment of Breastfeeding After Delivery: a Randomized Controlled Trial
Brief Title: Metoclopramide to Aid Establishment of Breastfeeding:a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Associate Professor Chong Yap Seng, National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NHG-SIG/05011
Record Dates: First submitted 2005-12-11; First posted 2005-12-13 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Breastfeeding
Keywords: A drug is administered to initiate breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Active Comparator): Mothers with pre-term deliveries will receive metoclopramide 10 mg three times a day for the first 7 days and 2 times a day for the 8th to 10th day, and once a day for the 11th to 12th day
  Interventions: Drug: Metoclopramide (Maxolon)
- B (Placebo Comparator): Mothers with pre-term deliveries will receive metoclopramide 10 mg 3 times a day, 2 times a day from 8th to 10th day and once a day from 11th to 12th day
  Interventions: Drug: placebo
- C (Active Comparator): Mothers with full term deliveries will receive 10 mg metoclopramide, 3 times a day for the first 7 days, 2 times a day from 8th to 10th day, and once a day for day 11 to 12
  Interventions: Drug: Metoclopramide (Maxolon)
- D (Placebo Comparator): Mothers with full term deliveries will receive the placebo 10 mg three times a day, for 7 days, and two times a day from day 8 to day 10, and once a day from 11th to 12th day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Metoclopramide (Maxolon) — Mothers will be given metoclopramide 10 mg 3 times a day for 7 days, 2 times a day from day 8 to 10 and once a day from 11th to 12th day
  Other Names: Maxalon
  Arms: A; C
Drug: placebo — placebo 10 mg
  Arms: B; D

SUMMARY:
Hypothesis: Early use of oral metoclopramide can hasten and improve the establishment of lactogenesis II in mothers after preterm and term deliveries.

The study hopes to show that metoclopramide can be effective to establish and sustain Lactogenesis II for both preterm and term infants.

DETAILED DESCRIPTION:
Hypothesis:

Early Use of oral metoclopramide can hasten and improve the establishment of lactogenesis II in mothers after preterm and term deliveries.

Metoclopramide(Maxolon) promotes lactation by antagonizing the release of dopamine in the central nervous system, thereby increasing prolactin levels, and thus inducing or augmenting breast milk levels. While Metoclopramide has commonly been used to augment breast milk production and relactation, its efficacy in helping to establish lactogenesis II has never been studied in a controlled clinical trial. If effective, it may become a valuable tool in aiding the successful establishment of breastfeeding, particularly in high risk groups such as mothers of preterm babies.

If shown to be an effective galactogogue, the use of metoclopramide provides an inexpensive and safe means of establishing and sustaining lactogenesis II, indirectly improving the degree and duration of breastfeeding practiced by mothers of both term and preterm infants.

The anticipated benefits are expected to be greatest for preterm infants and their mothers.

ELIGIBILITY:
Inclusion Criteria:

All pregnant women who intend to breastfeed, from 28 weeks to term, who have not met the exclusion criteria

Exclusion Criteria:

1. Patients who have epilepsy or on anti-seizure medications,
2. Patients who have a history of significant depression or are on antidepressant drugs
3. Patients who have pheochromocytoma or uncontrolled hypertension
4. Patients who have intestinal bleeding or obstruction
5. Patients who have a known allergy or prior reaction to metoclopramide, or any other contraindications to the use of metoclopramide
6. Patients who have diabetes and hyperprolactinaemia
7. Patients with HIV infection
8. Current pregnancy complicated by fetal congenital anomalies and multiple fetuses

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
successful initiation of lactation as determined by lactogenesis II markers | 7 days postpartum

SECONDARY OUTCOMES:
weight change in baby 7 days after birth | 14 days postpartum
breastfeeding status at 14 days, 6 weeks, 3 months and 6 months after delivery | 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Y S CHONG, MBBS, Principal Investigator — Dept. of O & G, National University Hospital; Y S CHAN, BSN, Principal Investigator — DEPT OF O & G, NATIONAL UNIVERSITY HOSPITAL
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Result] Cregan MD, De Mello TR, Kershaw D, McDougall K, Hartmann PE. Initiation of lactation in women after preterm delivery. Acta Obstet Gynecol Scand. 2002 Sep;81(9):870-7. doi: 10.1034/j.1600-0412.2002.810913.x. PMID 12225305
- [Derived] Foong SC, Tan ML, Foong WC, Marasco LA, Ho JJ, Ong JH. Oral galactagogues (natural therapies or drugs) for increasing breast milk production in mothers of non-hospitalised term infants. Cochrane Database Syst Rev. 2020 May 18;5(5):CD011505. doi: 10.1002/14651858.CD011505.pub2. PMID 32421208